CLINICAL TRIAL: NCT05217173
Title: Functional Ankle Recovery After a Telerehabilitation Program for Patients With Sprain in the First Level of Care, Controlled Clinical Trial and Cost-effectiveness Study
Brief Title: Effectiveness of a Telerehabilitation Program in Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Juan Figueroa-García, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2021-3609-037
Record Dates: First submitted 2021-12-31; First posted 2022-02-01 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Ankle Sprain; Ankle Sprain 1St Degree; Ankle Sprain 2Nd Degree
Keywords: ankle sprain; telerehabilitation; effectiveness
MeSH Terms: conditions — Ankle Injuries | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: A controlled, randomized, pragmatic, single-blind and parallel clinical trial will be conducted. The independent variable will be the type of intervention (tele-rehabilitation vs usual care).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the maneuver, the collaborator who will invite and enter the study subject cannot be blinded to the group assignment. Subsequent evaluations (weekly) where the response variables will be measured will be carried out by a different collaborator, who will be blinded from the group to which each study subject corresponds. The data analyst will remain blinded and will not know to which groups each study subject belongs. The circumstances that may unmask the data of the study subjects for both the evaluator and the data analyst, will be when the study subject is removed from the study for any reason.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Rehabilitation service that will be provided remotely through information and communication technologies. It will start within the first 72 hours of having started with the condition (ankle sprain); They will receive a rehabilitation program using a mobile application (through a digital platform course), which will contain previously recorded videos with exercises that will serve as a guide for rehabilitation activities. The duration of the program will be 30 minutes a day, 5 days a week for 4 weeks.
  The content of the rehabilitation program will consist of e modules: 1) Information module on the disease and self-care, 2) Exercise module (Stretching, strengthening and proprioception).
  Interventions: Other: telerehabilitation
- Control group (No Intervention): Care service that is carried out by the Family Physician. The medical care that the patient with an ankle sprain will carry out with the Family Physician of the assigned office; Medical care will consist of the approach that the Doctor considers appropriate for the patient. The follow-up and time of disability will be the responsibility of the Physician in question

INTERVENTIONS:
Other: telerehabilitation — It will start within the first 72 hours of having started with the condition (ankle sprain); They will receive a rehabilitation program using a mobile application (through a digital platform course), which will contain previously recorded videos with exercises that will serve as a guide for rehabilitation activities. The duration of the program will be 30 minutes a day, 5 days a week for 4 weeks
  Arms: Intervention group

SUMMARY:
Ankle sprain is the most common sprain. Their care entails a high cost due to the incapacity for work that it generates. An early and timely intervention for the treatment of ankle sprain reduces the days of disability and functional recovery is faster. Strategies must be generated to provide timely care in rehabilitation. Telerehabilitation is a viable option to partially solve this problem. The purpose of this study is evaluate the effectiveness of functional ankle recovery after a telerehabilitation program in patients with sprain in the first level of care. Material and method: Controlled clinical trial, 92 subjects with grade 1 and 2 ankle sprain will be included; they will be divided into two groups, with randomized allocation. One group will receive usual care (n = 41) for ankle sprain and another will receive regular care plus telerehabilitation (n = 41) through a digital platform course, it will consist of video and written instructions. Foot and Ankle Ability Measure (FAAM) will be measured at baseline and weekly, until completing 4 weeks. Group experience: The group is trained for the development of the contents and the rehabilitation program, with clinical experience in evaluation, treatment and rehabilitation of ankle sprain.

DETAILED DESCRIPTION:
Ankle sprain (AS) is a soft tissue injury caused by a forced twisting movement that exceeds the normal limits of the joint. This injury can range from minimal tissue distention to complete tissue rupture, it is manifested clinically by pain, edema, and functional limitation of the joint.

AS is the injury most related to physically active people, the worldwide incidence is estimated at 1 in every 10,000 people, it represents 15 to 20% of all sports injuries and most frequently affects young adults, its frequency has led it to be considered a benign condition, however, 20% of cases will develop complications.

After presenting a AS, the effects on health and costs of care are frequently underestimated by health personnel and the patient. The economic costs of your care are highly variable, they depend on the severity of the injury and the therapeutic strategy used; in most cases, it takes several days of disability for the injured limb to recover, causing absenteeism from work. Likewise, the frequency and variability with which the treatment of is selected can affect the recovery time and the quality of life of the patient.

The most important component of treatment for AS is rehabilitation, since it accelerates healing and return to desired activities, however, a large number of patients do not receive this therapeutic component adequately. Currently there are changes in the way of care for patients, largely due to the health contingency caused by Coronavirus disease 2019 (COVID-19), where social distance is a recommended action, for this reason, telemedicine is a strategy that can help the care of patients with conditions that require rehabilitation; therefore, some countries included digital practice within their health system.

When introducing a new therapeutic strategy, the economic and health effects, positive and negative, must be taken into account; cost-effectiveness studies are useful to know these effects. There are few cost-effectiveness studies for AS where telerehabilitation is compared with usual treatments at the first level of care. The evidence on measures of the effectiveness of Interventions through the telerehabilitation of AS is limited. The results also suggest that, in low- and middle-income countries, these pieces of evidence are even more limited. Some studies have shown that a distance intervention in orthopedic consultations is equal to or more cost-effective than standard consultations, where patients must attend a face-to-face consultation with the doctor.

What is known is that early rehabilitation as an optimized treatment for ankle sprain reduces treatment costs and reduces complications. However, the effectiveness of a telerehabilitation intervention for AS like the one proposed in this protocol is still unknown.

The research question is: what is the effectiveness in functional ankle recovery after a tele-rehabilitation program in patients with sprain in the first level of care, in a controlled and cost-effective clinical trial?

Our objective is: to evaluate the effectiveness in functional recovery of the ankle after a telerehabilitation program in patients with sprain grade 1-2 in the first level of care, in a controlled and cost-effectiveness clinical trial.

The investigators hypothesize: there will be the same or greater functional recovery of the ankle after a telerehabilitation program compared to the usual treatment in patients with sprain grade 1-2 in the first level of care.

Trial design: a controlled, randomized, pragmatic, single-blind and parallel clinical trial will be conducted. The independent variable will be the type of intervention (telerehabilitation vs usual care). The participants assigned to the telerehabilitation group will carry out a rehabilitation program using a mobile application, which will contain previously recorded videos with exercises that will serve as a guide for the rehabilitation activities. The duration of the program will be 30 minutes a day, 5 days a week for 4 weeks. The control group will be patients with usual care for ankle sprain, in the outpatient consultation of their medical care unit, they will receive instructions to follow from their doctors during the 4-week period.

The dependent variable will be the functionality perceived by the patient. A collaborator will perform the group assignment, the initial assessment of ankle functionality perceived by the patient and the induction to the use of the application on the cell phone in the case of patients assigned to the intervention group. Subsequent (weekly) evaluations of functional perception of the ankle will be carried out by another collaborator who will be blinded and will not know to which group the evaluated patient belongs.

The personnel who will invite and train patients to enter and use the telephone or internet application will be family medicine resident physicians.

Methods.

Scope of study: patients presenting in primary care for the diagnosis of AS grade 1 and 2.

Experimental group (Telerehabilitation Group): Intervention. Rehabilitation service that will be provided remotely through information and communication technologies. It will start within the first 72 hours of having started with the condition (ankle sprain); they will receive a rehabilitation program using a mobile application (through a digital platform course), which will contain previously recorded videos with exercises that will serve as a guide for rehabilitation activities. The duration of the program will be 30 minutes a day, 5 days a week for 4 weeks. The control group will be patients with usual care for ankle sprain, in the outpatient consultation of their medical care unit, they will receive instructions to follow from their doctors during the 4-week period.

The content of the rehabilitation program will consist of 2 modules: 1) Information module on the disease and self-care, 2) Exercise module (Stretching, strengthening and proprioception). The exercise program is based on the recommendations of national and international clinical practice guidelines. Additionally, the patient will be provided with a physical activity diary to assess adherence to treatment and the time the patient remains on the platform will be monitored.

Control Group: Regular medical attention by family doctor. Care service that is carried out by the family doctor. The medical care that the patient with an ankle sprain will carry out with the family doctor; medical care will consist of the approach that the doctor considers appropriate for the patient. The follow-up and time of disability will be the responsibility of the doctor in question.

Criteria for interrupting the assigned intervention:

* By request of the participant.
* Due to worsening of the condition.

Strategies to improve compliance with the intervention: a weekly reminder will be made by phone call to patients.

Interventions prohibited during the trial: perform other types of rehabilitation exercises that are not contemplated in the study.

Sample size: to calculate the sample size, a clinical difference is considered in the Foot and Ankle Ability Measure (FAAM) based on the Hoch's study, where rehabilitation is performed in patients with chronic ankle instability based on joint mobilization, considering a minimal clinically important difference for measure ankle function at 4 weeks, having a result prior to the rehabilitation intervention of 78.27 in the activities of daily living (ADL) of Foot and Ankle Ability Measure (FAAM) (Standard Deviation 12.62) and post-intervention of 87.3 (Standard Deviation 11.07), with a minimum detectable difference of 9.1 with a significance level of 5% and a power of 90%, performing a size calculation for the difference in paired means, with a consideration of estimated losses of 20%, so the sample size is 41 subjects per group.

Recruitment: patients with a grade 1 and 2 ankle sprain diagnosis who have attended the family medicine consultation at Family Medicine Unit will be identified. Identification will be carried out through the medical information and clinical file area of the Unit. Patients will be contacted by phone and will be scheduled the next day. The number of patients diagnosed with AS is sufficient and frequent in the Unit.

Allocation of interventions and blinding: it will be carried out by simple randomization; the randomization process will be carried out by an individual other than the one who will assign the groups. The randomization procedure will be generated with the Excel program; due to the nature of the intervention, the collaborator who will invite and enter the study subject cannot be blinded to the group assignment. Subsequent evaluations (weekly) where the response variables will be measured will be carried out by a different collaborator, who will be blinded from the group to which each study subject corresponds. The data analyst will remain blinded and will not know to which groups each study subject belongs. The circumstances that may unmask the data of the study subjects for both the evaluator and the data analyst, will be when the study subject is removed from the study for any reason.

Data collection methods: to ensure the quality of the data obtained, the evaluators (resident physicians) will receive training to know and master the clinical scales. The monitoring of the intervention will be supervised by the responsible researcher. The input of the data obtained will be examined twice before being entered into the data matrix to verify its congruence, this review will be carried out by a collaborating researcher, all those data that are not plausible or outside the established ranges of values, they will have to be corroborated. It is considered to make phone calls and send text messages via cell phone to remind patients to carry out the rehabilitation exercises, in this way, promote the retention of patients in the study and achieve complete follow-up to the rehabilitation program.

Data monitoring: the monitoring of the data will be carried out by the main researcher, who will not have contact with the study subjects, nor with the evaluators. Weekly, an intermediate analysis of the data obtained will be carried out by the main researcher, who will make the decision to end the study when the objectives are met.

Damage: the study subjects will have the opportunity to report any type of adverse or unforeseen effect at any time, the report, if spontaneous, can be made by telephone to the collaborators or the principal investigator. In addition, in the weekly evaluation, there will be the opportunity to express any type of adverse event secondary to the rehabilitation maneuver. In case of corroborating any adverse effect secondary to the intervention, timely attention to the treating physician will be managed.

Audit: the progress of the results will be audited by the project's tutorial committee every six months or when the project's tutor committee considers it. Progress in the results will be reported to the local ethics and institutional research committee every six months.

Ethics and dissemination: it has the approval of the Local Ethics and Research Committee of the Mexican Institute of Social Security.

Informed consent: informed consent will be obtained by the collaborators of the research project at the time of identifying and inviting the study subject, that is, it will not be obtained by the main researcher. The informed consent form is a document approved and granted by the Mexican Institute of Social Security, through the Ethics and Research Committee.

Confidentiality: the data will be collected by the collaborators of the research project. The data will be collected in a single database to which, initially, only collaborators will have access, later it will be shared with the main researcher for data monitoring. The data will be kept in a computer equipment to which only the main investigator has access, for no reason will it be shared with personnel outside the study in order to maintain the confidentiality of the data before, during and after the trial.

Data access: at the end of the trial, only researchers will be able to access the data. Collaborators will only know the final results.

Additional and post-study care: the patients who have participated in the trial are guaranteed care within the health institution, so that attention to any damage suffered by the trial, will be followed and care. No additional compensation is established.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiaries of the Mexican Institute of Social Security
* Patients with grade 1 and 2 ankle sprain, and are within the first 72 hours of presenting it
* Over 18 years of age and under 61 (this age group is susceptible to receiving monetary transfers for medical disability due to being of working age).
* Who have formal employment with susceptibility to receive medical disability.
* That they agree to participate in the study and sign the informed consent.
* With a diagnosis of ankle sprain for the first time.
* That they have and know how to use a cell phone or computer, as well as its use with the internet.

Exclusion Criteria:

* - With a history of previous ankle sprain.
* With time greater than 72 hours after starting with the ankle sprain.
* Patients with neurological disorders.
* Patients who cannot read or write.
* Retired patients.
* With leg or foot ulcers.
* Users of steroids administered orally or intravenously.
* Pre-existing and concomitant ankle arthritis or history of significant ipsilateral or contralateral lower extremity injury / condition, eg. lower extremity joint prostheses, or central or peripheral neurological disorders.
* Fibromyalgia
* Neuromuscular plaque disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Ankle functionality perceived by the patient with foot and ankle ability measure | Within the first 72 hours of starting with the ankle sprain (baseline measurement) and thereafter, every week (for 4 weeks), until one month after entering the study
  The Foot and Ankle Ability Measurement (FAAM) is a self-report outcome instrument developed to assess the physical function of individuals with foot and ankle-related impairments. It is a 29-item questionnaire divided into two subscales: 1) Activities of Daily Living (ADL) with 21 items and the Sports subscale with 8 items. Each item is rated on a 5-point Likert scale (4 to 0) from "no difficulty at all" to "unable to do". Total item scores, range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, were converted into percentage scores. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction and a lower score is indicative of decreased function. The FAAM is reliable (ADL: ICC=0.89; Sport: ICC=0.087), valid and responsive to change after intervention. This measurement will be made in both groups (intervention and control).
Days of incapacity for work indicated by the doctor | They will be quantified from the first day after presenting the ankle sprain, until completing 4 weeks after being admitted to the study.
  The days of incapacity for work indicated by the treating physician to the study subject will be quantified, since the patient presented the ankle sprain, until completing 4 weeks from their entry into the study. This data will be obtained from the patient's electronic clinical record. The quantification of days of incapacity for work will be taken into account in both groups (intervention and control).

SECONDARY OUTCOMES:
Weekly minutes allocated to rehabilitation activities | The quantification of minutes will be carried out from the beginning of the study, every week, for 4 weeks.
  All the study subjects of the intervention group, from the moment they enter the study, will undergo a weekly face-to-face interview, where they will be asked, how many minutes did they perform the rehabilitation exercises daily for a week? These data will be collected in a record sheet, which will be filled out every week until the 4 weeks of the intervention are completed.
Change in Visual Analog Scale | Within the first 72 hours of starting with the ankle sprain (baseline measurement) and thereafter, every week (for 4 weeks), until one month after entering the study
  Self-reported levels of acute ankle pain at rest, will be recorded using separate 10 cm visual analog scale. Each visual analog scale will be anchored on the left (0 cm) with 'no pain' and 'worst pain' on the right (10 cm). Participants will place a single handwritten mark at one point along the 10 cm line. The linear distance from the left end of the line to the participants mark will be measured using a standard ruler and recorded in centimeters. Therefore, a higher numerical value reflects greater levels of pain intensity. Excellent test-retest reliability has been reported for assessing acute pain using a VAS (ICC=0.97

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Medicina Familiar 21, Iztacalco, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tiemstra JD. Update on acute ankle sprains. Am Fam Physician. 2012 Jun 15;85(12):1170-6. PMID 22962897
- [Result] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. 2016 consensus statement of the International Ankle Consortium: prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1493-1495. doi: 10.1136/bjsports-2016-096188. Epub 2016 Jun 3. PMID 27259750
- [Result] Postle K, Pak D, Smith TO. Effectiveness of proprioceptive exercises for ankle ligament injury in adults: a systematic literature and meta-analysis. Man Ther. 2012 Aug;17(4):285-91. doi: 10.1016/j.math.2012.02.016. Epub 2012 Mar 27. PMID 22459604
- [Result] Herzog MM, Kerr ZY, Marshall SW, Wikstrom EA. Epidemiology of Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):603-610. doi: 10.4085/1062-6050-447-17. Epub 2019 May 28. PMID 31135209
- [Result] Mun JU, Cho HR, Sung YJ, Kang KN, Lee J, Joo Y, Kim YU. The role of the anterior talofibular ligament area as a morphological parameter of the chronic ankle sprain. J Orthop Sci. 2020 Mar;25(2):297-302. doi: 10.1016/j.jos.2019.05.001. Epub 2019 May 16. PMID 31104886
- [Result] Chen ET, Borg-Stein J, McInnis KC. Ankle Sprains: Evaluation, Rehabilitation, and Prevention. Curr Sports Med Rep. 2019 Jun;18(6):217-223. doi: 10.1249/JSR.0000000000000603. PMID 31385837
- [Result] Brison RJ, Day AG, Pelland L, Pickett W, Johnson AP, Aiken A, Pichora DR, Brouwer B. Effect of early supervised physiotherapy on recovery from acute ankle sprain: randomised controlled trial. BMJ. 2016 Nov 16;355:i5650. doi: 10.1136/bmj.i5650. PMID 27852621
- [Result] Bleakley CM, O'Connor SR, Tully MA, Rocke LG, Macauley DC, Bradbury I, Keegan S, McDonough SM. Effect of accelerated rehabilitation on function after ankle sprain: randomised controlled trial. BMJ. 2010 May 10;340:c1964. doi: 10.1136/bmj.c1964. PMID 20457737
- [Result] Bleakley CM, Taylor JB, Dischiavi SL, Doherty C, Delahunt E. Rehabilitation Exercises Reduce Reinjury Post Ankle Sprain, But the Content and Parameters of an Optimal Exercise Program Have Yet to Be Established: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2019 Jul;100(7):1367-1375. doi: 10.1016/j.apmr.2018.10.005. Epub 2018 Oct 26. PMID 30612980
- [Result] Vuurberg G, Hoorntje A, Wink LM, van der Doelen BFW, van den Bekerom MP, Dekker R, van Dijk CN, Krips R, Loogman MCM, Ridderikhof ML, Smithuis FF, Stufkens SAS, Verhagen EALM, de Bie RA, Kerkhoffs GMMJ. Diagnosis, treatment and prevention of ankle sprains: update of an evidence-based clinical guideline. Br J Sports Med. 2018 Aug;52(15):956. doi: 10.1136/bjsports-2017-098106. Epub 2018 Mar 7. PMID 29514819
- [Result] Bendahou M, Khiami F, Saidi K, Blanchard C, Scepi M, Riou B, Besch S, Hausfater P. Compression stockings in ankle sprain: a multicenter randomized study. Am J Emerg Med. 2014 Sep;32(9):1005-10. doi: 10.1016/j.ajem.2014.05.054. Epub 2014 Jun 12. PMID 25043629
- [Result] Kaminski TW, Hertel J, Amendola N, Docherty CL, Dolan MG, Hopkins JT, Nussbaum E, Poppy W, Richie D; National Athletic Trainers' Association. National Athletic Trainers' Association position statement: conservative management and prevention of ankle sprains in athletes. J Athl Train. 2013 Jul-Aug;48(4):528-45. doi: 10.4085/1062-6050-48.4.02. PMID 23855363
- [Result] Fong DT, Hong Y, Chan LK, Yung PS, Chan KM. A systematic review on ankle injury and ankle sprain in sports. Sports Med. 2007;37(1):73-94. doi: 10.2165/00007256-200737010-00006. PMID 17190537
- [Result] Doherty C, Delahunt E, Caulfield B, Hertel J, Ryan J, Bleakley C. The incidence and prevalence of ankle sprain injury: a systematic review and meta-analysis of prospective epidemiological studies. Sports Med. 2014 Jan;44(1):123-40. doi: 10.1007/s40279-013-0102-5. PMID 24105612
- [Result] Hubbard-Turner T. Lack of Medical Treatment From a Medical Professional After an Ankle Sprain. J Athl Train. 2019 Jun;54(6):671-675. doi: 10.4085/1062-6050-428-17. Epub 2019 May 22. PMID 31116568
- [Result] Wells B, Allen C, Deyle G, Croy T. MANAGEMENT OF ACUTE GRADE II LATERAL ANKLE SPRAINS WITH AN EMPHASIS ON LIGAMENT PROTECTION: A DESCRIPTIVE CASE SERIES. Int J Sports Phys Ther. 2019 Jun;14(3):445-458. doi: 10.26603/ijspt20190445. PMID 31681503
- [Result] Lazarou L, Kofotolis N, Pafis G, Kellis E. Effects of two proprioceptive training programs on ankle range of motion, pain, functional and balance performance in individuals with ankle sprain. J Back Musculoskelet Rehabil. 2018;31(3):437-446. doi: 10.3233/BMR-170836. PMID 28946541
- [Result] Kemler E, van de Port I, Backx F, van Dijk CN. A systematic review on the treatment of acute ankle sprain: brace versus other functional treatment types. Sports Med. 2011 Mar 1;41(3):185-97. doi: 10.2165/11584370-000000000-00000. PMID 21395362
- [Result] Cervera-Garvi P, Ortega-Avila AB, Morales-Asencio JM, Cervera-Marin JA, Martin RR, Gijon-Nogueron G. Cross-cultural adaptation and validation of Spanish version of The Foot and Ankle Ability Measures (FAAM-Sp). J Foot Ankle Res. 2017 Aug 22;10:39. doi: 10.1186/s13047-017-0221-6. eCollection 2017. PMID 28852426
- [Result] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Result] Eechaute C, Vaes P, Van Aerschot L, Asman S, Duquet W. The clinimetric qualities of patient-assessed instruments for measuring chronic ankle instability: a systematic review. BMC Musculoskelet Disord. 2007 Jan 18;8:6. doi: 10.1186/1471-2474-8-6. PMID 17233912
- [Result] Delahunt E, Bleakley CM, Bossard DS, Caulfield BM, Docherty CL, Doherty C, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Remus A, Verhagen E, Vicenzino BT, Wikstrom EA, Gribble PA. Clinical assessment of acute lateral ankle sprain injuries (ROAST): 2019 consensus statement and recommendations of the International Ankle Consortium. Br J Sports Med. 2018 Oct;52(20):1304-1310. doi: 10.1136/bjsports-2017-098885. Epub 2018 Jun 9. PMID 29886432
- [Result] Hoch MC, Andreatta RD, Mullineaux DR, English RA, Medina McKeon JM, Mattacola CG, McKeon PO. Two-week joint mobilization intervention improves self-reported function, range of motion, and dynamic balance in those with chronic ankle instability. J Orthop Res. 2012 Nov;30(11):1798-804. doi: 10.1002/jor.22150. Epub 2012 May 18. PMID 22610971
- [Result] Richmond T, Peterson C, Cason J, Billings M, Terrell EA, Lee ACW, Towey M, Parmanto B, Saptono A, Cohn ER, Brennan D. American Telemedicine Association's Principles for Delivering Telerehabilitation Services. Int J Telerehabil. 2017 Nov 20;9(2):63-68. doi: 10.5195/ijt.2017.6232. eCollection 2017 Fall. PMID 29238450
- [Result] Dantas LO, Barreto RPG, Ferreira CHJ. Digital physical therapy in the COVID-19 pandemic. Braz J Phys Ther. 2020 Sep-Oct;24(5):381-383. doi: 10.1016/j.bjpt.2020.04.006. Epub 2020 May 1. No abstract available. PMID 32387004
- [Result] Bartolo M, Intiso D, Lentino C, Sandrini G, Paolucci S, Zampolini M; Board of the Italian Society of Neurological Rehabilitation (SIRN). Urgent Measures for the Containment of the Coronavirus (Covid-19) Epidemic in the Neurorehabilitation/Rehabilitation Departments in the Phase of Maximum Expansion of the Epidemic. Front Neurol. 2020 Apr 30;11:423. doi: 10.3389/fneur.2020.00423. eCollection 2020. PMID 32425880
- [Result] Tenforde AS, Iaccarino MA, Borgstrom H, Hefner JE, Silver J, Ahmed M, Babu AN, Blauwet CA, Elson L, Eng C, Kotler D, Homer S, Makovitch S, McInnis KC, Vora A, Borg-Stein J. Telemedicine During COVID-19 for Outpatient Sports and Musculoskeletal Medicine Physicians. PM R. 2020 Sep;12(9):926-932. doi: 10.1002/pmrj.12422. Epub 2020 Jul 10. PMID 32424977
- [Result] Buvik A, Bergmo TS, Bugge E, Smaabrekke A, Wilsgaard T, Olsen JA. Cost-Effectiveness of Telemedicine in Remote Orthopedic Consultations: Randomized Controlled Trial. J Med Internet Res. 2019 Feb 19;21(2):e11330. doi: 10.2196/11330. PMID 30777845
- [Result] Fatoye F, Gebrye T, Fatoye C, Mbada CE, Olaoye MI, Odole AC, Dada O. The Clinical and Cost-Effectiveness of Telerehabilitation for People With Nonspecific Chronic Low Back Pain: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jun 24;8(6):e15375. doi: 10.2196/15375. PMID 32357128
- [Result] Van Reijen M, Vriend I, van Mechelen W, Verhagen EA. Preventing recurrent ankle sprains: Is the use of an App more cost-effective than a printed Booklet? Results of a RCT. Scand J Med Sci Sports. 2018 Feb;28(2):641-648. doi: 10.1111/sms.12915. Epub 2017 Jun 19. PMID 28543566
- See also: Journal of Family Medicine Andalusian from Spain — https://www.samfyc.es/wp-content/uploads/2018/07/v17n2.pdf
- See also: is a guide of clinical practice of Mexican Institute of Social Security — http://www.imss.gob.mx/sites/all/statics/guiasclinicas/034GER.pdf